CLINICAL TRIAL: NCT01070381
Title: Daily Disposable Toric Comparative Trial in Europe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-346-C-008
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2012-01

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

ARMS (2):
- nelfilcon A / ocufilcon D (Other): Nelfilcon A contact lenses worn first, with ocufilcon D contact lenses worn second. Both products worn bilaterally on a daily wear, daily disposable basis for one week each.
  Interventions: Device: nelfilcon A contact lens; Device: ocufilcon D contact lens
- ocufilcon D / nelfilcon A (Other): Ocufilcon D contact lenses worn first, with nelfilcon A contact lenses worn second. Both products worn bilaterally on a daily wear, daily disposable basis for one week each.
  Interventions: Device: nelfilcon A contact lens; Device: ocufilcon D contact lens

INTERVENTIONS:
Device: nelfilcon A contact lens — Commercially marketed, toric, soft contact lens for daily disposable wear
Device: ocufilcon D contact lens — Commercially marketed, toric, soft contact lens for daily disposable wear

SUMMARY:
The purpose of this study is to investigate the subjective and objective performance of two daily disposable lenses for wearers with astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Current soft contact lens wearers able to be fit with soft toric lenses in the protocol-specified parameters.
* Achieve 0.5 or better distance visual acuity in each eye at time of dispense.
* Achieve acceptable or optimal fit in each eye at time of dispense.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Habitual daily disposable contact lens wearer.
* Sleeps in contact lenses overnight.
* Currently enrolled in an ophthalmic clinical trial.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants were enrolled but not dispensed due to failing inclusion/exclusion criteria. These participants were included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Period: Period 1, 1 Week of Wear
Arm/Group | Nelfilcon A / Ocufilcon D | Ocufilcon D / Nelfilcon A
Started | 109 (One subject could not be dispensed into Period 1 product. Subject started Period 2 wear.) | 107
Completed | 109 (One subject could not continue into Period 2 due to product unavailability.) | 107
Not Completed | 0 | 0
Period: Period 2, 1 Week of Wear
Arm/Group | Nelfilcon A / Ocufilcon D | Ocufilcon D / Nelfilcon A
Started | 109 | 107
Completed | 108 | 106
Not Completed | 1 | 1
Not completed — Handling | 0 | 1
Not completed — Unacceptable Vision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This reporting group includes all enrolled and dispensed subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 66

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall Comfort, as interpreted and reported by the participant on a questionnaire as a single, retrospective evaluation of 1-week's wear time. Overall comfort is measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 1 week of wear
Population: Analysis conducted per protocol, with exclusions due to reasons such as, major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Nelfilcon A; Ocufilcon D: Commercially marketed, toric, soft contact lens for daily disposable wear
Arm/Group | Nelfilcon A | Ocufilcon D
Number analyzed (Participants) | 213 | 213
Units on a Scale | 7.6 (1.9) | 7.6 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial = 87 days. Individual exposure = 2 weeks (1 week per product)
Description: All enrolled and exposed participants. Common lens-related symptoms were collected at baseline. Any 3-grade change (1 or more symptoms) from baseline in frequency or severity was recorded as an adverse event. Frequency was collected on a 5-point scale, with 0=never and 4=always. Severity was collected on a 5-point scale, with 0=none and 4=severe.
Arm/Group | Nelfilcon A | Ocufilcon D
Serious Adverse Events (participants affected / at risk) | 0/217 | 0/216
Other Adverse Events (participants affected / at risk) | 16/217 | 27/216
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfilcon A (N=217) | Ocufilcon D (N=216)
3-grade change in symptoms (frequency and/or severity) from baseline (Eye disorders) | 16 (16) | 27 (35) — As collected on a questionnaire. Symptoms included 1 or more of the following: lens awareness, discomfort, blurred vision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.